CLINICAL TRIAL: NCT06616350
Title: Impact of EsTOCma on OCD Family Members
Acronym: esTOCma family
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Gemma García-Soriano, Assistant Professor of Psychology, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1276901_FAMILY
Record Dates: First submitted 2024-09-19; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
Keywords: stigma; obsessive-compulsive disorder; family; mental health literacy; esTOCma; app
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Social Stigma; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This study is a two-arm randomized controlled trial with measurements taken at two time points: pre-intervention and post-intervention. Participants who met the inclusion criteria were automatically randomized within the app into either the experimental or control group using a 1:1 allocation ratio. The experimental group received the intervention through the esTOCma app, and completed the assessment questionnaires before and after the intervention. Participants in the control group did not receive the intervention and completed the assessment questionnaires again 10 days after the pre-assessment (post-intervention).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Participants used the app esTOCma
  Interventions: Device: esTOCma: an app to fight stigma associated with OCD
- Control group (No Intervention): Participants did nothing

INTERVENTIONS:
Device: esTOCma: an app to fight stigma associated with OCD — The intervention consists of playing a serious game, called esTOCma, on a mobile phone. In the game, players must use their knowledge to battle the stigma monster of OCD, complete 10 missions, and release 10 individuals who have been afflicted by the esTOCma monster, a creature that feeds on false beliefs and misinformation in society.
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to test the acceptability, feasibility, and effectiveness of esTOCma in families and relatives of individuals with obsessive-compulsive disorder (OCD).

Specifically, a randomized controlled trial with two conditions (experimental and control) has been carried out in a sample of families and relatives of individuals with obsessive-compulsive disorder to assess pre-post-intervention changes. Researchers will compare experimental and control group to see if after using the app there is: lower stigma, higher knowledge and understanding about OCD, higher intention to seek help, and higher self-esteem and lower obsessive-compulsive symptoms. and there are no changes in the control group.

The experimental group received the intervention through the esTOCma app.

ELIGIBILITY:
Inclusion Criteria:

* having signed the informed consent
* being over 18 years of age;
* having an Android or iOS mobile device with Internet access
* being a family member of a person diagnosed with OCD.

Exclusion Criteria:

* not completing one or more of the evaluation time points (pre- or post-intervention)
* not finishing the intervention (experimental group only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change on mental health literacy about OCD | through study completion, an average of 10 days
  Score change on mental health literacy about OCD from baseline to after app completion in the experimental group, and no changes after 10 days in the control group. It will be assessed with the Mental Health Literacy Questionnaire (MHL) that was designed to assess level of knowledge about OCD, specifically the understanding of OCD and its treatment. Higher scores indicate higher knowledge.
Change in social distance | through study completion, an average of 10 days
  Score change in social distance from baseline to after app completion (experimental group), or no changes on the control group after 10 days. It will be assessed with the Social Distance Scale (SDS) that employs a four-point Likert scale, ranging from 0 to 3, to assess an individual's willingness to interact with a person who has a mental disorder as depicted in the assigned OC vignette across seven different settings. Higher scores indicate a stronger desire for social distance.
Change in stigma associated with OCD | through study completion, an average of 10 days
  Score change in stigma from baseline to app completion (estimation of 10 days) in the experimental group, and after 10 days in the control group. Stigma will be assessed by the Spanish version of the Attribution Questionnaire (AQ-27) that assesses public stigma related to a vignette. Respondents rate 27 items on a Likert-type scale from 1 to 9. Elevated scores indicate greater public stigma.
Change in help-seeking intention | through study completion, an average of 10 days
  Score change in help-seeking intention General after the intervention in the experimental group, and after 10 days in the control group. It will be assessed with the Help-Seeking Questionnaire (GHSQ) that comprises 10 items assessing the intention to seek help from various sources in the event of experiencing symptoms similar to those described in the assigned OC vignette. Higher scores indicate a greater tendency to seek help.

SECONDARY OUTCOMES:
Change in obsessive-compulsive symptoms | through study completion, an average of 10 days
  Score change in obsessive-compulsive symptoms after the intervention (experimental group) or after 10 days (control group). It will be assessed with the Obsessive-Compulsive Inventory-Revised (OCI-R), an 18-item self-report questionnaire designed to assess the severity of OC symptoms. Higher scores indicate a greater degree of distress associated with OC symptoms.
Change on self-esteem | through study completion, an average of 10 days
  Change on self-esteem is measured with the Single-Item Self-Esteem Scale, a single item that measures self-esteem, with higher scores reflecting greater self-esteem

OTHER OUTCOMES:
Level of acceptability | through study completion, an average of 10 days
  After using the app, the acceptability level will be measured with three multiple choice questiones developed ad-hoc. Higher scores indicated a higher level of acceptability of the application.
System usability level | through study completion, an average of 10 days
  The usability of the app will be assessed after using it. We sill use the System Usability Scale to assess the usability and user satisfaction of the technology application. Scores above 70 are indicative of good usability, with higher scores denoting superior usability.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma García-Soriano, PhD, Principal Investigator — Universitat de València
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Time Frame: It will be available for 3 months after the publication of the study.
Access Criteria: Data will be available in the repository ZENODO
URL: https://zenodo.org

REFERENCES:
- [Background] Garcia-Soriano G, Arnaez S, Chaves A, Del Valle G, Roncero M, Moritz S. Can an app increase health literacy and reduce the stigma associated with obsessive-compulsive disorder? A crossover randomized controlled trial. J Affect Disord. 2024 Apr 1;350:636-647. doi: 10.1016/j.jad.2024.01.168. Epub 2024 Jan 20. PMID 38253133
- See also: Link to download the app from Google Play — https://play.google.com/store/apps/details?id=app.estocma.com&amp;hl=es
- See also: Link to download the app for iOs — https://apps.apple.com/uy/app/estocma/id1604651647